CLINICAL TRIAL: NCT05290584
Title: Influence of Preschool Children's Fundamental Movement Skills, Physical Activity, and Physical Fitness on Executive Function: A Prospective Observation Study
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hong Kong Baptist University (Other)
Collaborators: Beijing Normal University (Other); National Fitness Research Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: HKBU19481772
Record Dates: First submitted 2022-02-24; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Preschool Children; Executive Function; Fundamental Movement Skills; Physical Activity; Physical Fitness
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background: Early childhood is the most critical and rapid period of complete and healthy physical and cognitive development in human life. Executive function appears in early childhood and develops rapidly through complex coaction between environment and developmental processes. The preschool period is also characterized by a rapid growth in fundamental movement skills, physical activity and physical fitness. The scientific research on the relationship between fundamental movement skills, physical activity, physical fitness and executive function in preschoolers remains to be explored.

Objective: The purpose of this study was to examine the cross-sectional relationship between fundamental movement skills, physical activity, physical fitness and executive function in preschool children while controlling for potential confounding variables, examine the prospective influence (independent and interactive role) of preschooler's fundamental movement skills, physical activity and physical fitness on executive function, observe the preschoolers' fundamental movement skills, physical activity, physical fitness and executive function changes with age, and investigate gender and age differences in preschoolers' fundamental movement skills, physical activity, physical fitness and executive function.

Method: The proposed study consists of two phases, phase 1 is a cross-sectional study. Five hundred and five children aged 3-5 years will be recruited. The Test of Gross Motor Development Third Edition (TGMD-3) was used to assess children's fundamental movement skills. Preschool children's physical activity was monitored by accelerometer ActiGraph GT3X-BT. Physical fitness was tested using handgrip, 4*10m shuttle run, 20m shuttle run, 30s sit-ups, sit and reach, and balance beam. Executive function was tested by computer-based tasks including animal stroop, safari training and stop signal task. Phase 2 is a 12-month follow-up study. In the phase 2, all children enrolled in the baseline study will be followed up, the measurements and contents of the follow-up are the same as the baseline instrument.

ELIGIBILITY:
Inclusion Criteria:

* aged 3-5 years
* normally developing children with corresponding cognitive ability to participate in the data collection
* without heart, lung, liver, kidney and other important organ diseases or any neurological disorders (e.g., intellectual disability or autism spectrum disorder) that prevent children from performing normal PA.

Exclusion Criteria:

* children with cognitive disability
* with heart, lung, liver, kidney and other important organ diseases or any neurological disorders (e.g., intellectual disability or autism spectrum disorder) that prevent children from performing normal PA.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children will be recruited from kindergartens in Zhuhai through the support of Zhuhai Early Childhood Education Association and United International College. These two organizations have cooperated with many local kindergartens, which can help to recruit preschoolers.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Estimated)
Dates: Start 2021-10-11 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of body mass index | through study completion, 12 months
  Weight (measured in kilograms) and height (measured in meters) will be combined to report body mass index in kg/m^2. Change of body mass index between baseline and follow-up test is assessed.
Change of fundamental movement skills | through study completion, 12 months
  The Test of Gross Motor Development: Third Edition (TGMD-3) will be used to assess children's fundamental movement skills. The TGMD-3 provides two subscale and an overall composite score. Change of fundamental movement skills between baseline and follow-up test is assessed.
Change of sedentary behavior time | through study completion, 12 months
  Physical activity level will be objectively monitored using a tri-axial accelerometer ActiGraph GT3X-BT and is analyzed with the ActiLife 6.13 data analysis software. Counts per minute are recorded.The activity with lower than 819 counts per minute is categorized as sedentary behaviors. Overall time in sedentary behavior in minute is recorded as sedentary behavior time. Change of sedentary behavior time between baseline and follow-up test is assessed.
Change of light physical activity time | through study completion, 12 months
  Physical activity level will be objectively monitored using a tri-axial accelerometer ActiGraph GT3X-BT and is analyzed with the ActiLife 6.13 data analysis software. Counts per minute are recorded. The activity with higher than 820 counts per minute but lower than 3907 counts per minute is categorized as light physical activity. Overall time in light physical activity in minute is recorded as light physical activity time. Change of light physical activity time between baseline and follow-up test is assessed.
Change of moderate-to-vigorous physical activity time | through study completion, 12 months
  Physical activity level will be objectively monitored using a tri-axial accelerometer ActiGraph GT3X-BT and is analyzed with the ActiLife 6.13 data analysis software. Counts per minute are recorded. The activity with higher than 3908 counts per minute is categorized as moderate-to-vigorous physical activity. Overall time in moderate-to-vigorous physical activity in minute is recorded as moderate-to-vigorous physical activity time. Change of moderate-to-vigorous physical activity time between baseline and post-intervention tests is assessed. Change of moderate-to-vigorous physical activity time between baseline and follow-up test is assessed.
Change of cardiorespiratory fitness | through study completion, 12 months
  A 20-meter shuttle run is used to assess cardiorespiratory fitness. During the test, participants run back and forth on two running tracks 20 meters apart at an initial speed of 8.0km/h, followed by an increase of 0.5km/h per minute. Using a compact disc (CD) to control the speed, which systematically increases during the test. During the test, participants run back and forth, based on the timing of a beep from the CD recorder. If the participant fails to pass the other end of the 20 meters distance before the beep (after two attempts), the test is terminated and the number of shuttle legs completed is recorded and converted to an estimate of aerobic capacity. As we work with preschoolers, the track will be marked and the children will be led by an adult so they can master the pace of the run. Change of cardiorespiratory fitness between baseline and follow-up test is assessed.
Change of flexibility | through study completion, 12 months
  Flexibility will be assessed by sit and reach. During the test, the participants sit barefoot on the mat, feet straight with heels together, toes separated naturally, and the sole of their feet on the tester plate. Then the participant is asked to slowly bend forward and use their arms to push the edge of a movable board as far as they can without bending knees. The test is repeated twice, and the maximum value is recorded. Change of flexibility between baseline and follow-up test is assessed.
Change of muscular endurance | through study completion, 12 months
  Sit ups will be used to assess the muscular endurance of the trunk. The participants lie on their back with knees bent and arms crossed on the other shoulder. They stand up, sit up, and return to the starting position. The assistant holds the child's feet. The number of lifts in 30 seconds performed correctly to the seated position is recorded.Change of muscular endurance between baseline and follow-up test is assessed.
Change of muscular strength | through study completion, 12 months
  Hand grip strength is a classic strength test with high safety, accuracy, and suitability for younger children. Muscle strength is measured using a WCS-100 electronic dynamometer (Shanghai Wanqing Electronics Co., LTD.). During the test, participants stand in a quiet environment, relaxed, with their arms hanging down naturally. They hold the dynamometer, adjust the grip distance, grasp the dynamometer once with maximum strength, and the value is recorded. The left and right hands are measured alternately for three times, and the maximum value is recorded. To allow for proper rest, the interval between the three tests should be at least 15 seconds. Change of muscular strength between baseline and follow-up test is assessed.
Change of balance | through study completion, 12 months
  Dynamic balance will be measured by the balance beam test. The participants will stand on the platform behind the starting line, face the balance beam (3 m long, 10 cm wide, and 30 cm high), and raise their arms horizontally. When participants hear the start command, they will move their feet to the finish line in turn. The tester will give orders on the front side of the participant, start the stopwatch at the same time when the participant starts, and follow the participant to the finish line. At the same time, the tester will pay attention to observe the movements of the participant to prevent accidents. When either tiptoe of the participant crosses the finish line, the tester stops the clock immediately. The test is repeated twice, and the best result is recorded. Change of balance between baseline and follow-up test is assessed.
Change of speed-agility | through study completion, 12 months
  Speed-agility will be assessed by the 4 × 10-meter shuttle run test. When the participants hear the start signal, they run and turn a 10-meter track as fast as they can to cover a distance of 40 meters. At the end of each section of the track, participants have to touch the hand of one of the testers who have crossed the limit with their feet and then go back at maximum speed. The participant will be given two tests with one to two minutes breaks in between. The best of two tests is recorded. Change of speed-agility between baseline and follow-up test is assessed.
Change of inhibitory control | through study completion, 12 months
  Animal Stroop task will be used to assess inhibitory control. The reaction time difference between conflict and congruent conditions reflects the ability to handle cognitive conflicts. Change of inhibitory control between baseline and follow-up test is assessed.
Change of cognitive flexibility | through study completion, 12 months
  Stop-signal task will measure the ability to inhibit response and control impulsivity. The mean stop-signal delay indicates the ability to inhibit portent responses. Change of cognitive flexibility between baseline and follow-up test is assessed.
Change of working memory | through study completion, 12 months
  Safari training task will measure working memory. There are 90 trials in total and the task takes about 8 minutes. Change of working memory between baseline and follow-up test is assessed.

SECONDARY OUTCOMES:
Demographics questionnaire | through study completion, 12 months
  Participant's background information (gender, age, gestational week, delivery mode, gestation, feeding mode, main caregivers), sleep, parental PA behaviors and attitudes, and family information (family economic status, parents' education level, family structure) are recorded.
Screen time | through study completion, 12 months
  Screen time will be measured by the Parents' Role in Establishing healthy Physical activity and Sedentary behavior habits study (PREPS) questionnaire developed. The weighted minutes per day for each variable are then summed to generate total screen time.
Sleep | through study completion, 12 months
  Sleep will be assessed with the Children's Sleep Habits Questionnaire (CSHQ). It contains 56 items, 52 of which are rated on a three-point Likert scale. Each question is asked in relation to the previous one week.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing Normal University - Hong Kong Baptist University United International College, Zhuhai, Guangdong
  - Hong Kong Baptist University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No